CLINICAL TRIAL: NCT04064528
Title: Effects of Age on Amino Acid Delivery to Tendon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Chad C. Carroll, Assistant Professor, Purdue University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 1904022075
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Aging
Keywords: amino acid; tendon; aging
MeSH Terms: interventions — Amino Acids

STUDY DESIGN:
Intervention Model Description: Young (21-30 years old) and older (60-75 years) adults will each receive an oral bolus of 10 g of essential amino acids.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young (Active Comparator): Young adults will be given a 10 g oral bolus of amino acids.
  Interventions: Dietary Supplement: Amino Acids
- Older Adults (Experimental): Older adults will be given a 10 g oral bolus of amino acids.
  Interventions: Dietary Supplement: Amino Acids

INTERVENTIONS:
Dietary Supplement: Amino Acids — 10 g bolus of essential amino acids

SUMMARY:
Dietary amino acid supplementation may provide an effective means to promote tendon injury recovery and enhance collagen synthesis. While most published research has been completed in animal models, research with young adults has shown that a leucine-rich whey isolate consumed during a chronic resistance training (RT) intervention resulted in greater gains (~60%) in tendon CSA when compared to placebo. Leucine-rich diets have also improved tendon collagen content in rodents. Further, in our preliminary work utilizing microdialysis, we demonstrate that oral consumption of a leucine-rich amino acid beverage increased delivery of amino acids to tendons in young adults (21-30 years). However, whether aging alters the delivery of amino acids to tendons after oral consumption has not be investigated. In order to optimize amino acid dosing for chronic interventional studies, we wish to determine if aging influences amino acid concentration in the peritendinous (space around the tendon) space after oral consumption.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* body mass index >35 kg•m-2, those on medications known to affect protein or collagen metabolism, e.g. acetaminophen, ibuprofen, or prescription cyclooxygenase inhibitors, previous history of tendinopathy, or diabetes.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Achilles Peritendinous Amino Acid Levels in young and older adults | 0-6 hours post consumption
  Concentrations of amino acids will be measured from around the Achilles tendon

CONTACTS AND LOCATIONS:
Overall Officials: Chad C Carroll, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States